CLINICAL TRIAL: NCT06690632
Title: WAter Preparation for Magnetic Resonance Enterography in Crohn's Disease
Brief Title: WAter Preparation in Crohn's Disease's Imagery
Acronym: WAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC31/24/0238
Record Dates: First submitted 2024-10-29; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease (CD)
Keywords: Crohn; bowel distension; MRE; oral contrast media; tolerability
MeSH Terms: conditions — Crohn Disease | interventions — mineral acids, trace elements, water, drug combination

STUDY DESIGN:
Intervention Model Description: Prospective monocentric interventional single-blinded study. Randomization with 1:1 ratio between water preparation and standard preparation after stratification on past bowel resection and structuring phenotype.
  The exams and distension scores will be determined by two radiologists (one expert and one trainee) blinded on patient allocation group. In case of disagreement, a third radiologist (expert) will be required.
Who Masked: Outcomes Assessor
Masking Description: The exams and distension scores will be determined by two radiologists (one expert and one trainee) blinded on patient allocation group. In case of disagreement, a third radiologist (expert) will be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WATER (Experimental): ingestion of 1.5L of water 30min prior MRE acquisition
  Interventions: Other: water preparation
- PEG (Active Comparator): ingestion of 1.5L of water diluted PEG 45 min prior MRE acquisition (standard protocol)
  Interventions: Other: polyethylene glycol preparation

INTERVENTIONS:
Other: water preparation — ingestion of 1.5L of water 30min prior MRE acquisition
  Arms: WATER
Other: polyethylene glycol preparation — ingestion of 1.5L of water diluted PEG 45 min prior MRE acquisition (standard protocol)
  Arms: PEG

SUMMARY:
The goal of this clinical trial is to compare distension quality and patient experience of water and polyethylene glycol preparation as oral contrast media in Magnetic Resonance Enterography (MRE) in patients with Crohn's disease.

Thus, the main question it aims to answer is:

Is water sufficient to interpret MRE from patients with Crohn's disease?

Researchers will compare the standard protocol (polyethylene glycol) with water as bowel distension agent to see if it is possible to obtain a satisfying global distension of small bowel.

Participants will undergo the same procedures as standard care adding questionnaires and replacing water as the bowel distension agent for the MRE for patient randomized into the experimental group.

DETAILED DESCRIPTION:
Magnetic Resonance Enterography (MRE) is a key tool for clinicians managing patients with Crohn's disease. This exam has a high performance in the diagnosis of complications and determination of healing rate after medical treatment. Small bowel distension with 1-1.5L of distension agent is mandatory to allow an accurate analysis of disease activity. Indeed, an insufficient distension can lead to false positive (thickened appearance of the collapsed digestive tract). Nowadays, there no consensus on the agent used for bowel distension (polyethylene glycol (PEG), lactulose, mannitol, sorbitol). The major limitation of those agent is their sides effects (e.g. diarrhea, gas bloating, vomiting) that decrease patient adherence to treatment. Some have suggested use of water as distension agent because of its price and its low side effect incidence. Yet its utilization has been limited by the fear of early absorption that may limit bowel analysis.

The aim of our study is to compare standard protocol (polyethylene glycol) with water as bowel distension agent in IBD patients requiring MRE on their ability to obtain a satisfying global distension of small bowel (on a previously validated scale).

Due to the side effects linked to the ingestion of 1.5L of distension agent and the impossibility of evaluating the tolerance of each contrast agent if 2 MREs are carried out on the same day, each the participant will benefit from an MRI using a single preparation modality (water or PEG).

To ensure comparability of the groups, patients will be randomized with 1:1 ratio after stratification on past bowel resection and structuring phenotype. The exams and distension scores will be determined by two radiologists (one expert and one trainee) blinded on patient allocation group. Regarding side effects, patient will fulfill several questionnaires after the exam and at 48h (end of follow-up).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Crohn's Disease,
* need for MRE (determined by patient's gastroenterologist)

Exclusion criteria:

* < 18 years old,
* inability to obtain an informed consent,
* patient under guardianship or curatorship, allergy to PEG,
* contraindication to MRE (pregnancy, pace maker, claustrophobia in particular), - contraindication to phloroglucinol administration (phenylcetonuria),
* contraindication to gadolinium administration (kidney failure with glomerular filtration rate < 30/mL/1.73m², pregnancy, allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Bowel distension | The day of the Magnetic Resonance Enterography (MRE), specifically during the imaging procedure : from ingestion of distension product to end of imaging, approximately 1 hour
  Proportion of patients with an overall small bowel distension over 2 on a validated scale (from 0=poor to 4=excellent)

SECONDARY OUTCOMES:
self evaluated Tolerability of symptoms | before MRE
  Patient's symptoms using a self-questionnaire.
  The questionnaire have 7 symptoms detailed and the patient indicates if the symptom is either :
  "Very bearable" "Moderately bearable" "Slightly bearable" "Not at all bearable" "I have not had this symptom"
self evaluated Tolerability of symptoms | right after MRE
  Patient's symptoms using a self-questionnaire.
  The questionnaire have 7 symptoms detailed and the patient indicates if the symptom is either :
  "Very bearable" "Moderately bearable" "Slightly bearable" "Not at all bearable" "I have not had this symptom"
self evaluated Tolerability of symptoms | 48 hour post MRE
  Patient's symptoms using a self-questionnaire.
  The questionnaire have 7 symptoms detailed and the patient indicates if the symptom is either :
  "Very bearable" "Moderately bearable" "Slightly bearable" "Not at all bearable" "I have not had this symptom"

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Toulouse, Toulouse, France